CLINICAL TRIAL: NCT03513250
Title: Efﬁcacy and Safety of Hyoscine-n-butylbromide for the Alleviation of Early Catheter-related Bladder Discomfort After Elective Cesarean Delivery: a Randomized Controlled Trial
Brief Title: Efﬁcacy of Hyoscine-n-butylbromide in Catheter-related Bladder Discomfort After Elective Cesarean Section.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, lecturer in obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: bladder discomfort
Record Dates: First submitted 2018-04-10; First posted 2018-05-01 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Catheter Related Bladder Discomfort
MeSH Terms: interventions — Butylscopolammonium Bromide; Control Groups

STUDY DESIGN:
Intervention Model Description: A prospective randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyoscine-n-butylbromide group (Experimental): one ampoule of 20 mg of hyoscine-n-butylbromide (Buscopan, 20mg/Ampoule, CID/Boehringer ) will be administered intravenously immediately before the end of the cesarean section.
  Interventions: Drug: hyoscine-n-butylbromide
- control group (Placebo Comparator): the same volume (1 ml) of normal saline intravenously immediately before the end of the cesarean section.
  Interventions: Drug: control group

INTERVENTIONS:
Drug: hyoscine-n-butylbromide — one ampoule of 20 mg of hyoscine-n-butylbromide (Buscopan, 20mg/Ampoule, CID/Boehringer ) will be administered intravenously immediately before the end of the cesarean section.
  Arms: hyoscine-n-butylbromide group
Drug: control group — an equal volume(1 ml ) of normal saline will be administered before the end of cesarean section.
  Other Names: saline group
  Arms: control group

SUMMARY:
a prospective, randomized, placebo-controlled study will be conducted to investigate whether hyoscine-n-butylbromide has preventive effects on early postoperative CRBD in patients with urinary catheters who will undergo elective cesarean sections.

DETAILED DESCRIPTION:
The insertion of a urinary catheter in a patient undergoing a surgical procedure as cesarean section may lead to catheter-related bladder discomfort with varying degrees of severity during the postoperative period. Catheter-related bladder discomfort (CRBD) symptoms associated with an indwelling urinary catheter are similar to overactive bladder symptoms such as discomfort in the suprapubic region, urinary urgency, frequency, burning sensation with or without urge incontinence. Hyoscine N-butyl bromide also known as scopolamine is a drug with anticholinergic effects which exerts its effects by inhibiting the acetylcholine effects in parasympathetic receptors of smooth muscle cells, secretory glands, and central nervous system. Hyoscine-n-butylbromide was reported to be effective for treatment of CRBD.

More preventive than therapeutic drugs for CRBD should be investigated to improve patient comfort in all surgery patients with a urinary catheter.

A prospective, randomized, placebo-controlled study will be conducted to investigate whether hyoscine-n-butylbromide has preventive effects on early postoperative CRBD in patients with urinary catheters who will undergo elective cesarean sections.

ELIGIBILITY:
Inclusion Criteria:

* Elective primary or repeat cesarean section at or more than 38 weeks of gestation scheduled to insert a Foley catheter in the operation site.

Exclusion Criteria:

* • Urinary infection (assessed clinically and by urinalysis of midstream sample of urine (MSSU) with chemical indicator strips or dipsticks).

  * Contraindications for general anesthesia.
  * Maternal bladder, urethral and renal disorders causing irritating voiding problems such as dysuria, urge and stress incontinence.
  * Obstructive voiding symptoms like incomplete emptying, straining and voiding difﬁculty before surgery.
  * Overactive bladder (frequency: more than three times during the night or more than eight times in 24 h).
  * Morbid obesity.
  * Disturbances of the central nervous system (epilepsy, patients receiving MAO inhibitor).
  * Hypertensive disorders and/ or systemic disease requiring particular patient care (for example, cardiac disease, nephritic disorders).
  * Chronic analgesic abuse.
  * Hepatic or psychiatric disease will be excluded from the study.
  * A history of hypersensitivity or contraindication to hyoscine-n-butylbromide.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
catheter related bladder discomfort(CRBD) measured by numerical rating scale(NRS). | one hour post-operatively.
  the incidence and severity of CRBD between the 2 groups will be assessed by the 11-point numerical rating scale which is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of her pain.The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
  CRBD will be defined as the presence of an urge to void or suprapubic discomfort with an NRS score of ≥3.

SECONDARY OUTCOMES:
catheter related bladder discomfort(CRBD) measured by numerical rating scale(NRS). | two hours postopeatively.
  the incidence and severity of CRBD between the 2 groups will be assessed by the 11-point numerical rating scale which is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of her pain.The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
catheter related bladder discomfort(CRBD) measured by numerical rating scale(NRS). | six hours postoperatively.
  numerical rating scale.
Postoperative nausea and vomiting | 6 hours postoperative
  Postoperative nausea and vomiting
dry mouth | 6 hours postoperative
  the patient says"My mouth is dry"
facial flushing | 6 hours postoperative
  My face is hot.
painkiller | Up to 6 hours after study drug administration
  the need for rescue analgesics

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, MD, Principal Investigator — Cairo University
Locations (1):
- Ahmed Ashour, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided